CLINICAL TRIAL: NCT01064375
Title: Assessment of Safety and Immunogenicity of Intradermal Electroporation of tetwtCEA DNA in Patients With Colorectal Cancer
Brief Title: Safety Study of DNA Vaccine Delivered by Intradermal Electroporation to Treat Colorectal Cancer
Acronym: El-porCEA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maria Liljefors (Other)
Collaborators: Karolinska Institutet (Other); Swedish Institute for Infectious Disease Control (Other); Cyto Pulse Sciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Maria Liljefors, MD, senior consultant, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: El-porCEA; 2009-009863-75 (EudraCT Number)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: DNA vaccine; Electroporation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CEA DNA prime (cohort I) (Experimental): 5 patients, tetwtCEA DNA intradermal delivery with electroporation, not previously vaccinated with CEA66 DNA. Electrical pulses applied to vaccination sites in skin using Derma Vax immediately after DNA administration. One dose of Cyclophosphamide (300 mg/m2) will be given i.v. three days before each vaccination with tetwtCEA DNA.
  Interventions: Biological: tetwtCEA DNA (wt CEA with tetanus toxoid Th epitope); Device: Derma Vax (electroporation device); Drug: Cyclophosphamide
- CEA DNA boost (cohort II) (Experimental): 10 patients, tetwtCEA DNA intradermal delivery with electroporation, previously vaccinated with CEA66 DNA.Electrical pulses applied to vaccination sites in skin using Derma Vax immediately after DNA administration.One dose of Cyclophosphamide (300 mg/m2) will be given i.v. three days before each vaccination with tetwtCEA DNA.
  Interventions: Biological: tetwtCEA DNA (wt CEA with tetanus toxoid Th epitope); Device: Derma Vax (electroporation device); Drug: Cyclophosphamide
- CEA DNA prime + GM-CSF (cohort III) (Experimental): 5 patients, tetwtCEA DNA intradermal delivery with electroporation + GM-CSF, not previously vaccinated with CEA66 DNA.Electrical pulses applied to vaccination sites in skin using Derma Vax immediately after DNA administration.One dose of Cyclophosphamide (300 mg/m2) will be given i.v. three days before each vaccination with tetwtCEA DNA.
  Interventions: Biological: tetwtCEA DNA (wt CEA with tetanus toxoid Th epitope); Device: Derma Vax (electroporation device); Biological: GM-CSF; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: tetwtCEA DNA (wt CEA with tetanus toxoid Th epitope) — Two vaccinations at week 0 and 12. Intradermal administration of 400ug DNA/dose with electroporation
  Other Names: GM-CSF; cyclophosphamide
Device: Derma Vax (electroporation device) — Electrical pulses applied to vaccination sites in skin using Derma Vax immediately after DNA administration
  Other Names: GM-CSF; cyclophosphamide
Biological: GM-CSF — GM-CSF will be given for 4 consecutive days starting the day before the vaccination as an intradermal/subcutaneous administration of 150 ug of GM-CSF
  Other Names: cyclophosphamide
  Arms: CEA DNA prime + GM-CSF (cohort III)
Drug: Cyclophosphamide — One intravenous dose of 300 mg/m2 will be given three days before each vaccination with tetwtCEA DNA
  Other Names: Sendoxan

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a CEA DNA immunisation approach in patients with colorectal cancer. The DNA plasmid, tetwtCEA, encodes wild type human CEA fused to a tetanus toxoid T helper epitope. The vaccine will be delivered using an intradermal electroporation device, Derma Vax (Cyto Pulse Sciences). The following will be assessed:

* The efficiency of priming immunological responses to CEA by intradermal administration of CEA DNA in combination with electroporation.
* The efficiency of boosting immunological responses to CEA by intradermal administration of CEA DNA in combination with electroporation in subjects already vaccinated with CEA DNA.
* GM-CSF will be administered to half of the subjects primed with CEA DNA in combination with electroporation and any possible adjuvant effects of GM-CSF will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed AJCC stage II or III colorectal cancer
* Resection of the primary tumour without evidence of remaining macroscopic disease
* Allowable standard chemotherapy or radiotherapy in AJCC stage III completed minimum 2 months prior study entry
* Patients recruited from vaccination with CEA66 plasmid DNA must have completed trial at 18 months if immune response is proven or proven to be non-immune responders in two consecutive immunoassays.
* Age >18 years
* Karnofsky performance >80%
* Life expectancy of greater than 6 months
* Normal organ and marrow function
* Normal thyroid function as measured by serum T3, T4 and TSH
* Normal echocardiogram regarding arrhythmias (chronic or treated atrial fibrillation allowed)
* No concurrent treatment (chemotherapy or biological) may be planned during protocol treatment
* Women or men of reproductive potential must agree to use adequate contraception prior to study entry and for up to 3 months after the last injection
* Ability to understand and the willingness to sign an informed consent document

Exclusion Criteria:

* Immunotherapy or systemic corticosteroids within 8 weeks prior to entering the study
* Chemotherapy or radiotherapy within 2 months prior to entering the study
* Known hypersensitivity to GM-CSF
* Previous splenectomy or radiation therapy of the spleen
* Pregnancy or nursing
* HIV seropositivity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic intracranial disease, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of severe neurological, cardiovascular, renal, hepatic, respiratory, bone marrow dysfunction, organ graft or autoimmune disease (treated or not)
* Concomitant medication with an anticoagulant (acetylsalicylic acid and low-molecular weight heparin in prophylactic dose allowed)
* Other malignancy, except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Cardiac demand pacemakers or surgically implanted defibrillators.
* Patients that has any metal implants in the area of the injection, (e.g. shoulder implant in the upper arm or shoulder girdle)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and immunogenicity of a DNA immunisation approach where tetwtCEA DNA will be administered in combination with electroporation. | Within 72 weeks after immunisation

SECONDARY OUTCOMES:
To assess the efficiency of boosting immunological responses to CEA by intradermal administration of tetwtCEA DNA in combination with electroporation in subjects already vaccinated with CEA DNA | Within 72 weeks after immunisation
To compare effects (safety and immunogenicity) of additional adjuvance with GM-CSF | Within 72 weeks after immunsation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Liljefors, MD, PhD, Principal Investigator — Department of Oncology, Karolinska University Hospital/Institute
Locations (1):
- Department of Oncology, Karolinska University Hospital, Stockholm, Sweden